CLINICAL TRIAL: NCT00514800
Title: Community Based Trial of Home Blood Pressure Monitoring With Nurse Led Support in Patients With Stroke or TIA Recently Discharged From Hospital
Brief Title: Home Blood Pressure Monitoring Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: St George's, University of London (Other)
Collaborators: The Stroke Association, United Kingdom (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 07.0002; TSA 2006/05
Record Dates: First submitted 2007-08-09; First posted 2007-08-10 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2007-08

CONDITIONS: Stroke; Ischemic Attack, Transient
Keywords: Home monitoring; Primary care; Hypertension; TIA
MeSH Terms: conditions — Stroke; Ischemic Attack, Transient; Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Patients will be given a home blood pressure monitor and taught how to use it and how to respond to the readings using a standardised protocol and blood pressure targets. The study nurse will follow up patients at home after a month with additional telephone support according to a defined protocol. Patients will consult their own GP for medication changes when above target.
  GPs will be sent information about the study design, current guidelines and interpretation of home blood pressure readings.
  Interventions: Behavioral: Intervention - a validated home BP monitor and support from the specialist nurse
- Control (Active Comparator)
  Interventions: Behavioral: Control - usual care (BP monitoring by their practice)

INTERVENTIONS:
Behavioral: Intervention - a validated home BP monitor and support from the specialist nurse
  Arms: Intervention
Behavioral: Control - usual care (BP monitoring by their practice) — Patients will not receive a blood pressure monitor and will continue with usual GP care for hypertension management.
  GPs will be sent information about the study design, current guidelines and interpretation of home blood pressure readings.
  Arms: Control

SUMMARY:
Design: Community based randomised trial with follow up after 12 months Participants: 360 patients admitted with stroke or TIA within the past 9 months will be recruited from the wards or outpatients and randomly allocated into two groups. All patients will be visited by the specialist nurse at home at baseline when she will measure their BP and administer a questionnaire. The questionnaire and BP will be repeated at 12 months follow-up by another researcher blind as to whether the patient is in intervention or control group.

Intervention: Intervention patients will be given a validated home BP monitor and support from the specialist nurse. Control patients will continue with usual care (BP monitoring by their practice).

Main outcome measures in both groups after 12months: 1.Change in systolic BP 2.Cost effectiveness: Incremental cost of the intervention to the NHS and incremental cost per quality adjusted life year gained.

Study hypothesis. Home blood pressure monitoring with nurse support wil lead to lower blood pressure after 12 months compared with usual GP care

DETAILED DESCRIPTION:
High blood pressure in patients with stroke increases the risk of recurrence but management in the community is often inadequate. Home blood pressure monitoring may increase patients' involvement in their care, increase compliance, and reduce the need for patients to attend their GP if blood pressure is adequately controlled. However the value of home monitoring to improve BP control is unclear and there is now a window of opportunity for evaluation before their use becomes widespread in the UK. Furthermore its use in stroke patients presents unique challenges relating to the consequent neurological disability.

ELIGIBILITY:
Inclusion Criteria:

* Stroke or TIA in last 9 months
* Blood pressure above 140/85 when measured more than 1 week after stroke or on anti hypertensive medication

Exclusion Criteria:

* Severe illness likely to dominate pattern of care
* Already using home blood pressure monitor
* Non-English speaking
* Severe cognitive impairment (AMTS<7)
* Known secondary hypertension

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2007-03; Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Reduction in systolic blood pressure taken by study team at home visit | 12 months

SECONDARY OUTCOMES:
Reduction in diastolic blood pressure taken by study team at home visit | 12 months
Reduction in SBP and DBP taken by study team at home visit | 6 months
Number of prescribed anti hypertensive medications Number of changes to anti hypertensive medication | 12 months
EQ-5D | 12 months
FEAR | 12 months
Incremental cost of the intervention to the NHS and cost per QALY | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Sally Kerry, MSc, Principal Investigator — St George's, University of London
Locations (3):
- United Kingdom (3):
  - St. George's Healthcare Trust, London, London
  - St. Helier NHS Trust, Carshalton, Surrey
  - Mayday University Hospital, Croydon, Surrey

REFERENCES:
- [Derived] Kerry SM, Markus HS, Khong TK, Cloud GC, Tulloch J, Coster D, Ibison J, Oakeshott P. Home blood pressure monitoring with nurse-led telephone support among patients with hypertension and a history of stroke: a community-based randomized controlled trial. CMAJ. 2013 Jan 8;185(1):23-31. doi: 10.1503/cmaj.120832. Epub 2012 Nov 5. PMID 23128283
- [Derived] Kerry S, Markus H, Khong T, Doshi R, Conroy R, Oakeshott P. Community based trial of home blood pressure monitoring with nurse-led telephone support in patients with stroke or transient ischaemic attack recently discharged from hospital. Trials. 2008 Mar 19;9:15. doi: 10.1186/1745-6215-9-15. PMID 18353175